CLINICAL TRIAL: NCT00046592
Title: Mechanisms of Disability in Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1185; R01HL071223 (NIH)
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Arterial Occlusive Diseases; Peripheral Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Arterial Occlusive Diseases; Peripheral Vascular Diseases

SUMMARY:
To determine the mechanisms by which atherosclerotic peripheral artery disease (PAD) causes functional impairment and to define the degree to which peripheral artery disease associated pathophysiologic findings change over time.

DETAILED DESCRIPTION:
BACKGROUND:

Research demonstrates that men and women with lower extremity peripheral arterial disease (PAD) have poorer functioning than men and women without PAD. Preliminary data also indicate that more severe PAD at baseline, as measured by the ankle brachial index (ABI), is associated with a greater incidence of functional loss. However, the pathophysiologic mechanisms in the lower extremities responsible for PAD-related functional impairment and functional loss are not well defined.

DESIGN NARRATIVE:

The study cohort will consist of 790 individuals identified from three Chicago-area medical centers, of whom 500 will have PAD. Participants will undergo a baseline and two annual follow-up visits. Pathophysiologic findings in the lower extremities refer to reduced muscle mass, reduced muscle quality, and reduced peripheral sensory and motor function. Quality of muscle tissue is defined as the ratio of muscle force to muscle mass. Muscle mass will be measured with Computed Tomography (CT). Peripheral nerve function will be determined using surface electroneurography (ENG). Lower extremity functional measures will consist of measures pertinent to functioning during daily living and include six minute walk distance, seven-day physical activity level (assessed by accelerometer), walking speed, balance tests, and lower extremity muscle power.

The cross-sectional study will test the hypotheses that a) chronic lower extremity arterial ischemia is associated with specific pathophysiologic findings in lower extremity muscle and nerve and that b) these ischemia-related pathophysiologic findings are associated with lower extremity functional limitation.The longitudinal study will test the hypotheses that a) greater baseline lower extremity arterial ischemia as measured by ABI is associated with greater progression of pathophysiologic findings over two year follow-up and that b) greater ischemia-related pathophysiologic findings in the legs at baseline is associated with greater functional decline over two year follow up. Results will be used to develop interventions designed to improve lower extremity functioning and prevent functional decline in persons with PAD.

ELIGIBILITY:
No eligibility criteria

Ages: 59 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott — Northwestern University Feinberg School of Medicine